CLINICAL TRIAL: NCT03489512
Title: Clinical Phase IV Comparison Trial for 2% Chlorhexidine Skin Asepsis +70% Alcohol Versus Aqueous Chlorhexidine (2%) for the Prevention of Catheter-related Bacteremia in Critical Patients: Preliminary Study
Brief Title: Comparison Trial for Chloraprep Versus Aqueous Chlorhexidine (2%) for the Prevention of Catheter-related Bacteremia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative issues
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHLORAPREP
Record Dates: First submitted 2018-03-14; First posted 2018-04-05 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-08

CONDITIONS: Sepsis Affecting Skin; Central Venous Catheter Related Bacteremia

STUDY DESIGN:
Intervention Model Description: Patients will receive one or the other treatment depending on where and when they are treated and will continue the treatment until the end.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Chloraprep) (Experimental): 2% chlorhexidine gluconate with 70% isopropyl alcohol with a sterile 3ml single dose applicator. Use for the preparation of the skin before insertion of the central venous catheters and at each dressing change.
  Interventions: Drug: A (Chloraprep)
- B (Clorhexidine 2%) (Active Comparator): 2% aqueous base chlorhexidine (10 ml single dose containers). Use for the preparation of the skin before insertion of the central venous catheters and at each dressing change.
  Interventions: Drug: B (Clorhexidine 2%)

INTERVENTIONS:
Drug: A (Chloraprep) — Chloraprep will be used for the insertion and maintenance of the intravascular device while it is in use (Chlorhexidine 2% + alcohol 70%)
  Other Names: Chloraprep
  Arms: A (Chloraprep)
Drug: B (Clorhexidine 2%) — Aqueous clorhexidine (2%) will be used for the insertion and maintenance of the intravascular device while it is in use
  Other Names: Clorhexidine 2%
  Arms: B (Clorhexidine 2%)

SUMMARY:
A multicentre, open-label clinical trial of two groups comparing cutaneous asepsis with chlorhexidine gluconate at 2% + isopropyl alcohol 70% in relation to the placement of central venous catheters (Study group) with standard asepsis with aqueous chlorhexidine at 2% (Group Control). The incidence of catheter related bacteremia, the incidence of colonization of the skin and the incidence of colonization of the central venous catheter will be evaluated.

DETAILED DESCRIPTION:
A multicentre, open-label clinical trial of two groups comparing cutaneous asepsis with chlorhexidine gluconate at 2% + isopropyl alcohol 70% in relation to the placement of central venous catheters (Study group) with standard asepsis with aqueous chlorhexidine at 2% (Group Control). The incidence of catheter related bacteremia, the incidence of colonization of the skin and the incidence of colonization of the central venous catheter will be evaluated.

The patients will assigned to the treatment group depending on where and when they are treated (site A or site B) and will continue the treatment until the end (continuous design): the patients of Site A will receive the first treatment option and those of Site B will receive the second treatment option during the first 6 months. After this, a rest period of 1 month will be established, during which patients will not be recruited and any of the two cutaneous aseptic methods will be used indiscriminately, in the opinion of the responsible nursing staff. After the resting period, the treatments will be reversed during the following 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU.
* Patients with age greater than or equal to 18 years.
* Patients who require at least one central venous catheters during 48h or more.
* Obtaining informed consent.

Exclusion Criteria:

* Intolerance or known allergy to chlorhexidine, isopropyl alcohol or orange yellow S (E110).
* High probability of death within 48 hours after admission.
* Use of coated catheter.
* Previously included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter-related bacteremia | Up to 48 hours after discharge from the ICU.
  Measure the effect of cutaneous asepsis with chlorhexidine gluconate 2% + isopropyl gluconate 70% on the incidence of catheter-related bacteremia in the critical patient with respect to the control group.

SECONDARY OUTCOMES:
Incidence of pericatheter skin colonization | Through study completion, an average of 1 year
  Measure the effect that cutaneous asepsis with chlorhexidine gluconate 2% + isopropyl 70% has on the incidence of pericatheter skin colonization with respect to the control group.
  Measure with a microbiological culture from the skin area
Incidence of colonization of the central venous catheter | Through study completion, an average of 1 year
  Measure the effect of cutaneous asepsis with chlorhexidine gluconate 2% + isopropyl 70% on the incidence of colonization of the central venous catheter with respect to the control group.
  Culture of the tip of the removed catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Ramirez Galleymore, Principal Investigator — Hospital La Fe